CLINICAL TRIAL: NCT05856123
Title: Single-site, Pilot Study Evaluating SimPull as a Primary Means of Lateral Patient Transfer
Brief Title: A Study to Evaluate SimPull for Lateral Patient Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: The Patient Company, LLC (Unknown)
Responsible Party: Principal Investigator, Deanna L. Covelli, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-004929
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-08

CONDITIONS: Lateral Patient Transfer
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group 1: Standard of Care Transfer (No Intervention): After cardiac catheterization lab or electrophysiology lab procedure, the subject will be moved from one bed to another using the current standard of practice lateral patient transfer methods by nursing staff.
- Group 2: SimPull Device Transfer (Experimental): After cardiac catheterization lab or electrophysiology lab procedure, the subject will be moved from one bed to another using the SimPull device.
  Interventions: Device: SimPull Lateral Transfer Device
- Group 3: Clinicians (Active Comparator): Study clinicians complete a survey after conducting intervention or standard of care on participants.
  Interventions: Other: Survey

INTERVENTIONS:
Device: SimPull Lateral Transfer Device — Automated lateral transfer device
  Arms: Group 2: SimPull Device Transfer
Other: Survey — Complete Survey
  Arms: Group 3: Clinicians

SUMMARY:
The purpose of this research is to test an investigational device called SimPull to see if it is a more efficient method of transferring a patient from one bed to another compared to that of current methods. The purpose of this research is to gather information on the safety and effectiveness of the SimPull device.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring lateral transfer for an invasive cardiac procedure to and from gurney to exam table.
* Patients requiring lateral transfer for an invasive cardiac procedure to and from exam table to gurney.
* Patient does not have compound fractures or cervical fractures present.
* Patient does not have skin damage or open wounds to the dorsal cavity.
* Patient or legally authorized representative (LAR) must be able/present to sign consent.

Exclusion Criteria:

* Patients who do not require lateral transfer for an invasive cardiac procedure to and from gurney to exam table.
* Patients who do not require lateral transfer for an invasive cardiac procedure to and from exam table to gurney.
* Patient has compound fractures or cervical fractures present.
* Patient has skin damage or open wounds to the dorsal cavity.
* Patient or legally authorized representative (LAR) are unable/present to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Covelli, MSN, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only Group 1 and Group 2 were actual participants who were enrolled in the study. Data was only collected for Group 1 and Group 2. Group 3 consisted of clinicians (provided the intervention or standard of care to Group 1 and Group 2 participants). Group 3 did not receive any intervention nor were they enrolled in the study. Group 3 only participated in the post intervention/standard of care survey.
Period: Overall Study
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer | Group 3: Clinicians
Started | 50 | 50 | 7
Completed | 50 | 50 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 3 was not enrolled in the study. They participated in the evaluation of this intervention as providers. This group did not receive the study intervention nor standard of care, and no demographic data was collected from this group. Only data from Group 1 and Group 2 is reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 34 | 67
  >=65 years | 17 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 37 | 33 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Lateral Transfer
Description: The average total time (minutes) it took to complete a lateral transfer.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer
Number analyzed (Participants) | 50 | 50
minutes | 33.40 (121.40) | 4.094 (1.688)

2. Primary Outcome: The Number of Staff Involved in a Transfer
Description: The average number of staff members engaged during transfers
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: staff members
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer
Number analyzed (Participants) | 50 | 50
staff members | 4.98 (0.87) | 4.92 (0.88)

3. Primary Outcome: Average Weight of Participants
Description: The average weight (kilograms) of participants who underwent a lateral transfer
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer
Number analyzed (Participants) | 50 | 50
kilograms | 86.24 (20.23) | 89.47 (22.57)

4. Secondary Outcome: Clinician Satisfaction
Description: Number of survey responses where clinicians indicated they were satisfied with the transfer method
Time Frame: Baseline
Population: A survey was provided to every study clinician who participated in a standard of care lateral transfer or a SimPull lateral transfer. A survey was provided to every study clinician who participated in a standard of care lateral transfer or a SimPull lateral transfer. There were 14 more survey responses in the SimPull group because some of the SimPull transfers required the involvement of more than one of the study clinicians to complete the transfer of the patient.
Measure: Count of Units; unit: Survey Responses
Units Other Than Participants: Survey Responses
Arm/Group | Group 3: Clinicians
Number analyzed (Participants) | 7
Number analyzed (Survey Responses) | 114
Survey Responses
  Standard of Care-subject moved using the standard of practice lateral patient transfer methods: number analyzed (Survey Responses) | 50
  Standard of Care-subject moved using the standard of practice lateral patient transfer methods | 44
  SimPull Device Transfer-subject moved using the SimPull automated lateral transfer device: number analyzed (Survey Responses) | 64
  SimPull Device Transfer-subject moved using the SimPull automated lateral transfer device | 40

5. Secondary Outcome: The Number of Survey Responses From Clinicians Who Indicated They Were Very Likely to Experience Injury During Transfers
Description: Measured by a post transfer survey where clinicians indicated how likely they feel they are to be injured during lateral patient transfer using standard transfer methods versus SimPull on a scale of "Not at all likely", "Not likely", "Neutral", "Likely", or "Very Likely."
Time Frame: Baseline
Population: A survey was provided to every study clinician who participated in a standard of care lateral transfer or a SimPull lateral transfer. There were 14 more survey responses in the SimPull group because some of the SimPull transfers required the involvement of more than one of the study clinicians to complete the transfer of the patient.
Measure: Count of Units; unit: Survey Responses
Units Other Than Participants: Survey Responses
Arm/Group | Group 3: Clinicians
Number analyzed (Participants) | 7
Number analyzed (Survey Responses) | 114
Survey Responses
  Standard of Care-subject moved using the standard of practice lateral patient transfer methods: number analyzed (Survey Responses) | 50
  Standard of Care-subject moved using the standard of practice lateral patient transfer methods | 0
  SimPull Device Transfer-subject moved using the SimPull automated lateral transfer device: number analyzed (Survey Responses) | 64
  SimPull Device Transfer-subject moved using the SimPull automated lateral transfer device | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 1 hour.
Description: CTCAE version 5.0. Group 3 did not participate in the intervention or standard of care and were not enrolled in the study. Adverse events were not collected from the clinician participants in Group 3.
Groups:
- Group 3: Clinicians: Group 3 participants were not enrolled to the study and participated only in study evaluation.
Arm/Group | Group 1: Standard of Care Transfer | Group 2: SimPull Device Transfer | Group 3: Clinicians
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/0
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT05856123/Prot_SAP_000.pdf